CLINICAL TRIAL: NCT03194711
Title: Bioabsorbable Drug-eluting Scaffolds (BVS)-Optical Coherence Tomography (OCT) Imaging Study
Brief Title: BVS-OCT Imaging Study
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 16-2757
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Coronary Disease
Keywords: Percutaneous Coronary Revascularization; Optical Coherence Tomography; Stents, Drug-Eluting
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stable CAD
  Interventions: Device: BVS implantation

INTERVENTIONS:
Device: BVS implantation — BVS implantation using conventional semicompliant or non-compliant balloon

SUMMARY:
The single center retrospective study evaluates the acute and long term outcomes of bioabsorbable drug-eluting scaffolds (BVS) implantation in 50 consecutive coronary artery disease (CAD) patients using optical coherence tomography (OCT) imaging.

DETAILED DESCRIPTION:
I. INTRODUCTION Bioabsorbable drug-eluting scaffolds ("BVS") have emerged as a potential major breakthrough for treatment of coronary artery lesions providing a possibility to overcome the long term limitations of conventional stent implantation which precludes future surgical revascularization, eliminates reactive vasomotion, impairs noninvasive imaging and exposes patients to the risk of very late stent thrombosis. BVS have been extensively studied in clinical trials. Treatment of noncomplex obstructive coronary artery disease with BVS was within the prespecified margin for noninferiority compared to Xience stent with respect to target lesion failure at 1 year in the latest large-scale randomized trial (ABRORB III). Although the concept of self-degrading stent is attractive and the results from clinical trials have been promising, there is a paucity of data regarding the use of BVS in "real world" patients undergoing percutaneous intervention ("PCI"). The outcomes from a large BVS registry of patients with relatively unselected clinical characteristics and lesions were comparable to those reported for the second generation drug eluting stents ("DES"), however, the scaffold thrombosis rate in the first 30 days after implantation resembled that of the first generation DES suggesting that the lesion selection and procedure optimization require further improvement. BVS development has required new imaging modalities, assessment methodologies, and treatment strategies because their design, degradation rate, coating, changes in mechanical properties may affect safety and efficacy of the device. Due to its high resolution, Optical Coherence Tomography ("OCT") imaging has played a central role in understanding the short and long term performance of bioresorbable scaffolds.

II. STUDY AIM To evaluate the acute and long term outcomes of BVS implantation in consecutive coronary artery disease ("CAD") patients using OCT imaging.

III. STUDY POPULATION Fifty (50) consecutive patients who underwent PCI with BVS implantation and OCT imaging for treatment of CAD.

IV. STUDY DESIGN This is a single center retrospective analysis of data collected under the EXEMPT database (GCO# 02-0178) at the Cardiac Catheterization Laboratory at Mt. Sinai Hospital.

V. STUDY PROCEDURES Patients with stable CAD who underwent PCI with BVS implantation. Lesions were treated with pre-dilatation using conventional semicompliant or non-compliant balloon. The use of additional devices, cutting balloons or rotablator, were performed at the operator's discretion. The operator made the decision on BVS length and size. First OCT pullback (OCT-PRE) was performed before BVS implantation to analyze lesion stenosis, references, and plaque morphology including the extent and location of calcification. In addition, online co-registration of OCT with coronary angiogram was performed to confirm the correct spatial orientation of OCT findings. The second OCT pullback (OCT - POST) was performed after BVS implantation followed by post-dilatation (20 atm). Angio-OCT co-registration was used to assess acute post-procedural results.

VI. STUDY OUTCOMES

* Acute lumen gain after BVS implantation by quantitative coronary angiography ("QCA") and OCT; effect of coronary calcification on lumen gain, BVS apposition and expansion.
* Review of the clinical follow up data which was collected at 1 month and 12 months after the procedure

VII. IMAGE ANALYSIS

QCA analysis. In each patient, the treated segment (in-scaffold) and the peri-scaffold segment (defined as 5 mm proximal and distal to the scaffold edge) will be analyzed by QCA in paired matched angiographic views before and after procedure using metallic markers at the proximal and distal ends of the device. Minimal lumen diameter (MLD), reference vessel diameter, percentage of area stenosis, and lesion length will be measured by two experienced analysts using dedicated software (QCA-QAngioXA 7.3; Medis) as previously described. Acute lumenal gain will be defined as the difference between MLD immediately after procedure and MLD before BVS implantation. In addition, the presence of angiographic calcification will be assessed. Calcification will be identified by angiography as readily apparent radiopacities within the vascular wall at the site of stenosis and will be classified as none/mild or moderate (radiopacities noted only during the cardiac cycle before contrast injection)/severe (radiopacities visible without cardiac motion before contrast injection usually compromising both sides of the lumen).

OCT lesion analysis will be performed offline at 1-mm interval according to previously validated criteria and as we previously described. The minimal and reference lumen diameter and area will be measured to calculate percent lumen area stenosis. Plaques will be classified as fibrous, lipid, or calcified. For each lipid plaque, the maximal lipid arc will be measured at 1-mm interval and the minimal thickness of the fibrous cap will be assessed. The degree of circumferential extent of calcification will be quantified at 1 mm interval by measuring the maximal calcification arc.

OCT analysis of BVS will be performed at 1-mm interval within the entire stented segment and at 5 mm proximal and distal to the BVS edge. For each cross section analyzed, the area, mean, minimal and maximal diameters of the BVS will be measured automatically with manual corrections if appropriate. The proximal and distal reference vessel area (RVA) will be calculated as the mean of the largest two lumenal areas 5 mm distal and proximal to the BVS edge. Acute strut fracture will be suspected if isolated struts are detected lying unopposed in the lumen with no connection to other surrounding stent struts. 3D OCT reconstruction with QAngio OCT RE software (Medis) will be performed to confirm the diagnosis. Incomplete strut apposition (ISA) will be defined as the presence of struts separated from the underlying vessel wall. The percentage of ISA will be calculated as a ratio of malapposed struts number to the total number of struts observed at 1-mm interval. Since abluminal border of the struts can be visualized in BVS, we will assess the ISA area for each frame with malapposed struts. The percentage of Residual Area Stenosis (RAS) will be calculated as: [(1 - (minimal lumen area/RVA))] ×50 ; the eccentricity index as the ratio between the minimal and the maximal diameter. The symmetry index will be defined as (maximal stent diameter - minimal stent diameter)/(maximal stent diameter). OCT analysis will be performed in Mount Sinai Cath Lab Core imaging laboratory.

VIII. PROPENSITY-MATCHED COMPARISON BETWEEN BVS AND DES A retrospective analysis will be performed on 50 study patients who underwent PCI with BVS and consecutive patients who underwent DES implantation in Mount Sinai catheterization laboratory with the comparator sample size of 50. The DES patients will be selected from the Mount Sinai imaging database. Propensity score matching will be performed to reduce the effect of confounding factors in the retrospective study for two groups of patients with different recruitment periods. Multiple logistic regression analysis will include the following variables as covariates: previous MI, previous CABG, CAD family history, history of smoking, dyslipidemia, diabetes mellitus, use of atherectomy device, stent/BVS post-dilatation, stent/BVS diameter and length, maximal calcium arc by OCT and total number of treated vessels.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who underwent PCI with BVS implantation and OCT imaging for treatment of CAD

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mount Sinai Catheterization laboratory patients who who underwent PCI with BVS implantation and OCT imaging for treatment of CAD
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Acute lumen gain by quantitative coronary angiography (QCA) | 1 year
  Acute lumen gain after BVS implantation by quantitative coronary angiography (QCA)
Acute lumen gain by Optical Coherence Tomography (OCT) | 1 year
  Acute lumen gain after BVS implantation by OCT

SECONDARY OUTCOMES:
Major adverse cardiac events | 1 year
  Major adverse cardiac events, defined as a composite of cardiac death, myocardial infarction, and target lesion

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, MRCP, FACC, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mattesini A, Secco GG, Dall'Ara G, Ghione M, Rama-Merchan JC, Lupi A, Viceconte N, Lindsay AC, De Silva R, Foin N, Naganuma T, Valente S, Colombo A, Di Mario C. ABSORB biodegradable stents versus second-generation metal stents: a comparison study of 100 complex lesions treated under OCT guidance. JACC Cardiovasc Interv. 2014 Jul;7(7):741-50. doi: 10.1016/j.jcin.2014.01.165. PMID 25060016
- [Background] Serruys PW, Onuma Y, Garcia-Garcia HM, Muramatsu T, van Geuns RJ, de Bruyne B, Dudek D, Thuesen L, Smits PC, Chevalier B, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Hebert KM, Rapoza R, Ormiston JA. Dynamics of vessel wall changes following the implantation of the absorb everolimus-eluting bioresorbable vascular scaffold: a multi-imaging modality study at 6, 12, 24 and 36 months. EuroIntervention. 2014 Mar 20;9(11):1271-84. doi: 10.4244/EIJV9I11A217. PMID 24291783
- [Background] Serruys PW, Chevalier B, Dudek D, Cequier A, Carrie D, Iniguez A, Dominici M, van der Schaaf RJ, Haude M, Wasungu L, Veldhof S, Peng L, Staehr P, Grundeken MJ, Ishibashi Y, Garcia-Garcia HM, Onuma Y. A bioresorbable everolimus-eluting scaffold versus a metallic everolimus-eluting stent for ischaemic heart disease caused by de-novo native coronary artery lesions (ABSORB II): an interim 1-year analysis of clinical and procedural secondary outcomes from a randomised controlled trial. Lancet. 2015 Jan 3;385(9962):43-54. doi: 10.1016/S0140-6736(14)61455-0. Epub 2014 Sep 14. PMID 25230593
- [Background] Kimura T, Kozuma K, Tanabe K, Nakamura S, Yamane M, Muramatsu T, Saito S, Yajima J, Hagiwara N, Mitsudo K, Popma JJ, Serruys PW, Onuma Y, Ying S, Cao S, Staehr P, Cheong WF, Kusano H, Stone GW; ABSORB Japan Investigators. A randomized trial evaluating everolimus-eluting Absorb bioresorbable scaffolds vs. everolimus-eluting metallic stents in patients with coronary artery disease: ABSORB Japan. Eur Heart J. 2015 Dec 14;36(47):3332-42. doi: 10.1093/eurheartj/ehv435. Epub 2015 Sep 1. PMID 26330419
- [Background] Ellis SG, Kereiakes DJ, Metzger DC, Caputo RP, Rizik DG, Teirstein PS, Litt MR, Kini A, Kabour A, Marx SO, Popma JJ, McGreevy R, Zhang Z, Simonton C, Stone GW; ABSORB III Investigators. Everolimus-Eluting Bioresorbable Scaffolds for Coronary Artery Disease. N Engl J Med. 2015 Nov 12;373(20):1905-15. doi: 10.1056/NEJMoa1509038. Epub 2015 Oct 12. PMID 26457558
- [Background] Capodanno D, Gori T, Nef H, Latib A, Mehilli J, Lesiak M, Caramanno G, Naber C, Di Mario C, Colombo A, Capranzano P, Wiebe J, Araszkiewicz A, Geraci S, Pyxaras S, Mattesini A, Naganuma T, Munzel T, Tamburino C. Percutaneous coronary intervention with everolimus-eluting bioresorbable vascular scaffolds in routine clinical practice: early and midterm outcomes from the European multicentre GHOST-EU registry. EuroIntervention. 2015 Feb;10(10):1144-53. doi: 10.4244/EIJY14M07_11. PMID 25042421
- [Background] Garcia-Garcia HM, Serruys PW, Campos CM, Muramatsu T, Nakatani S, Zhang YJ, Onuma Y, Stone GW. Assessing bioresorbable coronary devices: methods and parameters. JACC Cardiovasc Imaging. 2014 Nov;7(11):1130-48. doi: 10.1016/j.jcmg.2014.06.018. Epub 2014 Nov 10. PMID 25459595
- [Background] Ormiston JA, Serruys PW, Onuma Y, van Geuns RJ, de Bruyne B, Dudek D, Thuesen L, Smits PC, Chevalier B, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Hebert KM, Rapoza R, Garcia-Garcia HM. First serial assessment at 6 months and 2 years of the second generation of absorb everolimus-eluting bioresorbable vascular scaffold: a multi-imaging modality study. Circ Cardiovasc Interv. 2012 Oct;5(5):620-32. doi: 10.1161/CIRCINTERVENTIONS.112.971549. Epub 2012 Oct 9. PMID 23048057
- [Background] Kini AS, Vengrenyuk Y, Pena J, Motoyama S, Feig JE, Meelu OA, Rajamanickam A, Bhat AM, Panwar S, Baber U, Sharma SK. Optical coherence tomography assessment of the mechanistic effects of rotational and orbital atherectomy in severely calcified coronary lesions. Catheter Cardiovasc Interv. 2015 Nov 15;86(6):1024-32. doi: 10.1002/ccd.26000. Epub 2015 May 11. PMID 25964009
- [Background] Kini AS, Motoyama S, Vengrenyuk Y, Feig JE, Pena J, Baber U, Bhat AM, Moreno P, Kovacic JC, Narula J, Sharma SK. Multimodality Intravascular Imaging to Predict Periprocedural Myocardial Infarction During Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2015 Jun;8(7):937-45. doi: 10.1016/j.jcin.2015.03.016. PMID 26088511
- [Background] Tearney GJ, Regar E, Akasaka T, Adriaenssens T, Barlis P, Bezerra HG, Bouma B, Bruining N, Cho JM, Chowdhary S, Costa MA, de Silva R, Dijkstra J, Di Mario C, Dudek D, Falk E, Feldman MD, Fitzgerald P, Garcia-Garcia HM, Gonzalo N, Granada JF, Guagliumi G, Holm NR, Honda Y, Ikeno F, Kawasaki M, Kochman J, Koltowski L, Kubo T, Kume T, Kyono H, Lam CC, Lamouche G, Lee DP, Leon MB, Maehara A, Manfrini O, Mintz GS, Mizuno K, Morel MA, Nadkarni S, Okura H, Otake H, Pietrasik A, Prati F, Raber L, Radu MD, Rieber J, Riga M, Rollins A, Rosenberg M, Sirbu V, Serruys PW, Shimada K, Shinke T, Shite J, Siegel E, Sonoda S, Suter M, Takarada S, Tanaka A, Terashima M, Thim T, Uemura S, Ughi GJ, van Beusekom HM, van der Steen AF, van Es GA, van Soest G, Virmani R, Waxman S, Weissman NJ, Weisz G; International Working Group for Intravascular Optical Coherence Tomography (IWG-IVOCT). Consensus standards for acquisition, measurement, and reporting of intravascular optical coherence tomography studies: a report from the International Working Group for Intravascular Optical Coherence Tomography Standardization and Validation. J Am Coll Cardiol. 2012 Mar 20;59(12):1058-72. doi: 10.1016/j.jacc.2011.09.079. Erratum In: J Am Coll Cardiol. 2012 May 1;59(18):1662. Dudeck, Darius [corrected to Dudek, Darius]; Falk, Erlin [corrected to Falk, Erling]; Garcia, Hector [corrected to Garcia-Garcia, Hector M]; Sonada, Shinjo [corrected to Sonoda, Shinjo]; Troels, Thim [corrected to Thim, Troels]; van Es, Gerrit-Ann [correct. PMID 22421299